CLINICAL TRIAL: NCT01296932
Title: A Phase I, Open, Dose Escalation Trial With BI 836826 in Patients With Advanced Chronic Lymphocytic Leukaemia
Brief Title: BI836826 Dose Escalation in Relapsed Chronic Lymphocytic Leukaemia (CLL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1270.1; 2010-021488-34 (EudraCT Number)
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — BI 836826

ARMS (1):
- Patients with relapsed CLL (Experimental): Patients with relapsed CLL after at least two prior treatment regimens will receive BI 836826.
  Interventions: Drug: BI 836826

INTERVENTIONS:
Drug: BI 836826 — Monotherapy with BI 836826 at escalating dose levels administered as an intravenous infusion.

SUMMARY:
Adult patients with chronic lymphocytic leukaemia who experience a relapse after at least two prior treatment regimens may be enrolled in this trial. The trial will examine whether monotherapy with BI 836826 is safe and tolerable at escalating dose levels.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of relapsed or refractory chronic lymphocytic leukaemia.
2. At least two prior treatment regimens for chronic lymphocytic leukaemia.
3. At least one criterion for active disease as defined by the International Workshop on CLL.
4. Absolute lymphocyte count lower than 200 x 10^9/l .
5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1 or 2.
6. Age 18 years or older.
7. Written informed consent which is consistent with International Conference on Harmonisation - Good Clinical Practice (ICH-GCP) guidelines and local legislation.

Exclusion criteria:

1. Treatment with anti Cluster of Differentiation (CD) 20 therapy within 4 weeks, or alemtuzumab within 8 weeks, or any cytotoxic antileukemia therapy within 2 weeks, Ibrutinib or Idelalisib within 1 week prior to the first administration of the trial drug.
2. Prior allogeneic stem cell transplantation.
3. Active autoimmune haemolytic anemia.
4. Active autoimmune thrombocytopenia.
5. Known transformation to an aggressive B-cell malignancy.
6. Concurrent treatment with relevant doses of systemic glucocorticosteroids.
7. Prior history of malignancy other than chronic lymphocytic leukaemia (exceptions to this rule are defined in the clinical trial protocol).
8. Aspartate aminotransferase or alanine aminotransferase > 2.5 x upper limit of normal.
9. Total bilirubin > 1.5 x upper limit of normal.
10. Absolute Neutrophil Count < 1.000/µl.
11. Platelets < 25.000/µL.
12. Estimated Glomerular Filtration Rate <45 mL/min.
13. Proteinuria Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or higher.
14. Significant concurrent disease.
15. Any infectious disease requiring treatment at the time of enrolment or within the previous 2 weeks.
16. Hepatitis B or C.
17. Human Immunodeficiency Virus (HIV) infection.
18. Cytomegalovirus (CMV) viremia.
19. Women of childbearing potential not using a highly effective method of birth control during the trial until one year after the last dose.
20. Pregnancy or breast feeding.
21. Known or suspected active alcohol or drug abuse.
22. Treatment with another investigational drug within the past four weeks before start of therapy or concomitantly with this trial.
23. Prior treatment with BI 836826.
24. Patients unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-02-11 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (10):
- Belgium (3):
  - Brussels - UNIV Saint-Luc, Brussels
  - Edegem - UNIV UZ Antwerpen, Edegem
  - UNIV UZ Gent, Ghent
- France (3):
  - INS Paoli-Calmettes, Marseille
  - CTR Investigation Clinique, onco, Montpellier, Montpellier
  - INS Universitaire du Cancer, Toulouse
- Germany (4):
  - Universitätsklinikum Köln (AöR), Cologne
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Ulm, Ulm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase-1,single arm,open-label,dose escalation trial, patients with advanced chronic lymphocytic leukemia. While the first part of the trial was still in progress, recruitment was ended by the sponsor before the maximum tolerated dose(MTD) or Optimal Biological Dose(OBD) was reached.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites to ensure that all patients met all inclusion/exclusion criteria. Patients were not to be entered to trial treatment if any one of the specific entry criteria were not met.
Groups:
- BI 836826 1 Milligram: Patients were administered BI 836826-1 milligram solution for infusion after dilution intravenously as one single dose within a 14-day cycle
- BI 836826 3 Milligram: Patients were administered BI 836826-3 milligram solution for infusion after dilution intravenously as one single dose within a 14-day cycle
- BI 836826 9 Milligram: Patients were administered BI 836826-9 milligram solution for infusion after dilution intravenously as one or two doses within the first cycle followed by single doses within all following 14-day cycles
- BI 836826 25 Milligram: Patients were administered BI 836826-25 milligram solution for infusion after dilution intravenously as two doses within the first cycle followed by single doses within all following 14-day cycles
- BI 836826 50 Milligram: Patients were administered BI 836826-50 milligram solution for infusion after dilution intravenously as two doses within the first cycle followed by single doses within all following 14-day cycles
- BI 836826 100 Milligram: Patients were administered BI 836826-100 milligram solution for infusion after dilution intravenously as two doses within the first cycle followed by single doses within all following 14-day cycles
- BI 836826 200 Milligram: Patients were administered BI 836826-200 milligram solution for infusion after dilution intravenously as two doses within the first cycle followed by single doses within all following 14-day cycles
- BI 836826 400 Milligram: Patients were administered BI 836826-400 milligram solution for infusion after dilution intravenously as two doses within the first cycle followed by single doses within all following 14-day cycles
- BI 836826 800 Milligram: Patients were administered BI 836826-800 milligram solution for infusion after dilution intravenously as two doses within the first cycle followed by single doses within all following 14-day cycles
Period: Overall Study
Arm/Group | BI 836826 1 Milligram | BI 836826 3 Milligram | BI 836826 9 Milligram | BI 836826 25 Milligram | BI 836826 50 Milligram | BI 836826 100 Milligram | BI 836826 200 Milligram | BI 836826 400 Milligram | BI 836826 800 Milligram
Started | 3 | 3 | 6 | 6 | 3 | 3 | 6 | 3 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 3 | 3 | 6 | 6 | 3 | 3 | 6 | 2 | 4
Not completed — Dose limiting toxicity | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Progressive disease | 2 | 0 | 1 | 1 | 2 | 3 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1
Not completed — Investigator decision | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Not completed — No clinical benefit anymore | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — IV problems, administration not possible | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — per protocol | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Low benefit and too many side effects | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — No adequate treatment response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Dosage already reduced, AE still present | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All patients who received at least one application of the drug BI 836826.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 836826 1 Milligram | BI 836826 3 Milligram | BI 836826 9 Milligram | BI 836826 25 Milligram | BI 836826 50 Milligram | BI 836826 100 Milligram | BI 836826 200 Milligram | BI 836826 400 Milligram | BI 836826 800 Milligram | Total
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 3 | 3 | 6 | 3 | 4 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.7 (8.4) | 74.3 (5.7) | 63.3 (10.0) | 58.7 (9.6) | 63.3 (13.2) | 61.0 (17.0) | 73.3 (5.4) | 70.7 (11.4) | 69.5 (6.5) | 66.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 0 | 1 | 1 | 4 | 0 | 1 | 11
  Male | 1 | 2 | 5 | 6 | 2 | 2 | 2 | 3 | 3 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity data were not collected for the study. Race was not collected in France due to law (These are the missing/unknown).
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    White | 3 | 2 | 4 | 2 | 1 | 2 | 2 | 3 | 2 | 21
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 2 | 4 | 2 | 1 | 4 | 0 | 2 | 16

OUTCOME MEASURES:

1. Secondary Outcome: Best Percentage Change From Baseline in Number of Lymphocytes in the Peripheral Blood
Description: In most patients with relapsed or refractory chronic lymphocytic leukaemia (CLL), malignant B-cells represent the majority of lymphocytes in the peripheral blood. Reduction of CLL-cells was assessed in the peripheral blood by absolute lymphocyte count, and flow cytometry. The number of lymphocytes in the peripheral blood was analysed in terms of the best percentage change from baseline until start of subsequent CLL therapy or progressive disease (PD).
Time Frame: baseline and ≥8 day after a completed infusion of a cycle and before Chronic Lymphocytic Leukemia (CLL) therapy; data collected up to cut-off date 26Oct2016, Up to 1809 days
Population: All patients who received at least one application of the drug BI 836826, had a baseline and at least one post-baseline assessment of the number of lymphocytes in the peripheral blood.
Measure: Mean (Standard Deviation); unit: Percentage of change (%)
Arm/Group | BI 836826 1 Milligram | BI 836826 3 Milligram | BI 836826 9 Milligram | BI 836826 25 Milligram | BI 836826 50 Milligram | BI 836826 100 Milligram | BI 836826 200 Milligram | BI 836826 400 Milligram | BI 836826 800 Milligram
Number analyzed (Participants) | 3 | 3 | 6 | 5 | 3 | 3 | 6 | 3 | 4
Percentage of change (%) | -11.39 (31.39) | -21.20 (10.08) | -48.21 (57.39) | -48.15 (34.01) | -49.35 (31.44) | -81.81 (11.03) | -79.22 (39.94) | -93.40 (9.76) | -47.14 (103.29)

2. Secondary Outcome: Number of Patients With Improved Haemoglobin Count for at Least Two Subsequent Response Assessments
Description: In patients with haemoglobin counts below the limits of normal at baseline, improvement in this count during therapy potentially indicated a benefit for the patient. Number of patients with improved haemoglobin count for at least two subsequent response assessments which fulfil International Workshop on Chronic Lymphocytic Leukemia (IWCLL) response criteria for Complete Remission (CR) or Partial Remission (PR). The response was assessed before Progressive Disease (PD) or start of new Chronic Lymphocytic Leukaemia (CLL) therapy.
Time Frame: ≥8 day after a completed infusion of a cycle and before Chronic Lymphocytic Leukemia (CLL) therapy; data collected up to cut-off date 26Oct2016, Up to 1809 days
Population: Treated Set (TS): All patients who received at least one application of the drug BI 836826.
Measure: Count of Participants; unit: Participants
Arm/Group | BI 836826 1 Milligram | BI 836826 3 Milligram | BI 836826 9 Milligram | BI 836826 25 Milligram | BI 836826 50 Milligram | BI 836826 100 Milligram | BI 836826 200 Milligram | BI 836826 400 Milligram | BI 836826 800 Milligram
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 3 | 3 | 6 | 3 | 4
Participants
  NO | 3 | 2 | 3 | 4 | 2 | 1 | 2 | 1 | 4
  YES | 0 | 1 | 3 | 2 | 1 | 2 | 4 | 2 | 0

3. Secondary Outcome: Number of Patients With Improved Platelet Count for at Least Two Subsequent Response Assessments
Description: In patients with platelet counts below the limits of normal at baseline, improvement in this count during therapy potentially indicated a benefit for the patient. Number of patients with improved platelet count for at least two subsequent response assessments which fulfil International Workshop on Chronic Lymphocytic Leukemia (IWCLL) response criteria for Complete Remission (CR) or Partial Remission (PR). The response was assessed before Progressive Disease (PD) or start of new Chronic Lymphocytic Leukaemia (CLL) therapy.
Time Frame: as for outcome 2
Population: TS
Measure: Count of Participants; unit: Participants
Arm/Group | BI 836826 1 Milligram | BI 836826 3 Milligram | BI 836826 9 Milligram | BI 836826 25 Milligram | BI 836826 50 Milligram | BI 836826 100 Milligram | BI 836826 200 Milligram | BI 836826 400 Milligram | BI 836826 800 Milligram
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 3 | 3 | 6 | 3 | 4
Participants
  NO | 2 | 2 | 2 | 3 | 3 | 1 | 3 | 0 | 3
  YES | 1 | 1 | 4 | 3 | 0 | 2 | 3 | 3 | 1

4. Secondary Outcome: Number of Patients With Improved Neutrophil Count for at Least Two Subsequent Response Assessments
Description: In patients with neutrophil count below the limits of normal at baseline, improvement in this count during therapy potentially indicated a benefit for the patient. Number of patients with improved neutrophil count for at least two subsequent response assessments which fulfil International Workshop on Chronic Lymphocytic Leukemia (IWCLL) response criteria for Complete Remission (CR) or Partial Remission (PR). The response was assessed before Progressive Disease (PD) or start of new Chronic Lymphocytic Leukaemia (CLL) therapy.
Time Frame: as for outcome 2
Population: TS
Measure: Count of Participants; unit: Participants
Arm/Group | BI 836826 1 Milligram | BI 836826 3 Milligram | BI 836826 9 Milligram | BI 836826 25 Milligram | BI 836826 50 Milligram | BI 836826 100 Milligram | BI 836826 200 Milligram | BI 836826 400 Milligram | BI 836826 800 Milligram
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 3 | 3 | 6 | 3 | 4
Participants
  YES | 1 | 3 | 5 | 4 | 1 | 2 | 5 | 3 | 1
  NO | 2 | 0 | 1 | 2 | 2 | 1 | 1 | 0 | 3

5. Secondary Outcome: Best Overall Response According to 'International Workshop on Chronic Lymphocytic Leukemia' (IWCLL) Criteria
Description: Response was assessed according to the IWCLL (International Workshop on Chronic Lymphocytic Leukemia) guidelines based on laboratory data from the peripheral blood and clinical examination by the investigator after each cycle prior to administration of the next dose of BI 836826, at the end of the treatment (EOT) visit, and at all Follow-up Visits. Best overall response will be analysed descriptively. Frequency distributions will be used to examine this endpoint.
Time Frame: Data collected up to cut-off date 26Oct2016 until Progressive disease (PD) to start of next Chronic Lymphocytic Leukaemia (CLL) therapy, Up to 1809 days.
Population: TS
Measure: Count of Participants; unit: Participants
Arm/Group | BI 836826 1 Milligram | BI 836826 3 Milligram | BI 836826 9 Milligram | BI 836826 25 Milligram | BI 836826 50 Milligram | BI 836826 100 Milligram | BI 836826 200 Milligram | BI 836826 400 Milligram | BI 836826 800 Milligram
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 3 | 3 | 6 | 3 | 4
Participants
  Complete remission | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Complete remission with incomplete marrow recovery | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial remission | 0 | 0 | 4 | 1 | 0 | 0 | 4 | 2 | 2
  Stable disease | 3 | 3 | 2 | 4 | 3 | 3 | 2 | 1 | 2
  Progressive disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not evaluable | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time from the first administration of BI 836826 until disease progression or death, whichever occurred first. Disease progression= At least one of the following:
  * 50+% increase in blood lymphocytes over baseline with an absolute number of B-lymphocytes of at least 5x109/L
  * Progression of lymphadenopathy
  * 50+% increase in the previously noted enlargement of the liver or new appearance of hepatomegaly
  * 50+% increase in the previously noted enlargement of the spleen or new appearance of splenomegaly
  * 50+% Decrease of platelet counts or to less than 100x109/L secondary to CLL and unrelated to autoimmune cytopenia
  * Decrease of haemoglobin levels by more than 20 g/L, or to less than 100 g/L secondary to CLL and unrelated to autoimmune cytopenia T Transformation to a more aggressive histology, e.g. Richter syndrome.
Time Frame: Data collected up to cut-off date 26Oct2016, Up to 1809 days.
Population: TS
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | BI 836826 1 Milligram | BI 836826 3 Milligram | BI 836826 9 Milligram | BI 836826 25 Milligram | BI 836826 50 Milligram | BI 836826 100 Milligram | BI 836826 200 Milligram | BI 836826 400 Milligram | BI 836826 800 Milligram
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 3 | 3 | 6 | 3 | 4
Days | 57.0 [15.0 to 316.0] | 86.0 [59.0 to 141.0] | 133.5 [79.0 to 281.0] | 81.0 [29.0 to 134.0] | 85.0 [16.0 to 106.0] | 114.0 [44.0 to 133.0] | 196.5 [98.0 to 247.0] | 113.0 [106.0 to 799.0] | 68.0 [51.0 to 74.0]

7. Secondary Outcome: Failure-free Survival
Description: Failure-free survival (FFS) was defined as the time from the first administration of BI 836826 until disease progression or death, or start of next Chronic Lymphocytic Leukemia (CLL) therapy, whichever occurred first. Disease progression= At least one of the following:
  * 50+% increase in blood lymphocytes over baseline with an absolute number of B-lymphocytes of at least 5x109/L
  * Progression of lymphadenopathy
  * 50+% increase in the previously noted enlargement of the liver or new appearance of hepatomegaly
  * 50+% increase in the previously noted enlargement of the spleen or new appearance of splenomegaly
  * 50+% Decrease of platelet counts or to less than 100x109/L secondary to CLL and unrelated to autoimmune cytopenia
  * Decrease of haemoglobin levels by more than 20 g/L, or to less than 100 g/L secondary to CLL and unrelated to autoimmune cytopenia T Transformation to a more aggressive histology, e.g. Richter syndrome.
Time Frame: Data collected up to cut-off date 26Oct2016, Up to 1809 days.
Population: TS
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | BI 836826 1 Milligram | BI 836826 3 Milligram | BI 836826 9 Milligram | BI 836826 25 Milligram | BI 836826 50 Milligram | BI 836826 100 Milligram | BI 836826 200 Milligram | BI 836826 400 Milligram | BI 836826 800 Milligram
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 3 | 3 | 6 | 3 | 4
Days | 57.0 [29.0 to 316.0] | 106.0 [59.0 to 141.0] | 152.5 [85.0 to 281.0] | 81.0 [29.0 to 134.0] | 85.0 [25.0 to 106.0] | 114.0 [54.0 to 133.0] | 196.5 [127.0 to 247.0] | 149.0 [120.0 to 799.0] | 100.0 [68.0 to 141.5]

8. Primary Outcome: Number of Patients With Dose-Limiting Toxicities Adverse Events (DLTs)
Description: Dose-Limiting Toxicities (DLTs) were defined as any drug-related non-haematologic adverse event of Common Terminology Criteria for AE (CTCAE) Grade 3 or higher, except infusion related reactions associated with the administration of BI 836826. In addition complications due to haematologic AEs were considered as DLTs and were added in more detail in an amendment later on.
Time Frame: 14 days after first administration of BI836826 (MTD evaluation period)
Population: The maximum tolerated dose (MTD) evaluation set: This includes all patients who were documented to have received at least one dose of trial medication and were not replaced for the MTD evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | BI 836826 1 Milligram | BI 836826 3 Milligram | BI 836826 9 Milligram | BI 836826 25 Milligram | BI 836826 50 Milligram | BI 836826 100 Milligram | BI 836826 200 Milligram | BI 836826 400 Milligram | BI 836826 800 Milligram
Number analyzed (Participants) | 3 | 3 | 6 | 5 | 3 | 3 | 6 | 3 | 3
Participants
  Total with dose limiting toxicities adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

9. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The maximum tolerated dose (MTD) was defined as the highest dose of BI 836826 studied for which the incidence of DLT was no more than 17% (i.e. 1 out of 6 patients) during the first treatment cycle. For those patients who received more than 1 cycle of BI 836826, all AEs corresponding to the DLT were considered for the purpose of confirming the MTD and for the selection of the recommended dose for treatment of the expansion cohort and for further development. All DLTs, occurring during the first or repeated treatment cycle were reported as significant AEs. As it was not possible to recruit a sufficient number of patients whilst the first part of the trial was still in progress, the recruitment was ended by the sponsor before the MTD or optimal biological dose (OBD) was reached.
Time Frame: 14 days after first administration of BI836826 (MTD evaluation period)
Population: The trial was discontinued prematurely due to lack of recruitment before the MTD based on the frequency of patients with DLTs in the first treatment cycle was reached.
Groups:
- BI 836826: Patients were administered BI 836826 solution for infusion after dilution intravenously as one or two doses within the first cycle followed by a single doses within all following 14-day cycles in the higher dose groups (>9 milligram BI 836826).
Arm/Group | BI 836826
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study medication until 6 weeks after last administration of BI 836826, up to 136 weeks
Description: The Treated set (TS) was used for adverse event reporting. (TS: This patient set consists of all patients who received at least one application of the BI drug BI 836826.)
Arm/Group | BI 836826 1 Milligram | BI 836826 3 Milligram | BI 836826 9 Milligram | BI 836826 25 Milligram | BI 836826 50 Milligram | BI 836826 100 Milligram | BI 836826 200 Milligram | BI 836826 400 Milligram | BI 836826 800 Milligram
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/6 | 0/3 | 0/3 | 0/6 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 4/6 | 3/6 | 1/3 | 1/3 | 5/6 | 1/3 | 2/4
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 6/6 | 3/3 | 3/3 | 6/6 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 836826 1 Milligram (N=3) | BI 836826 3 Milligram (N=3) | BI 836826 9 Milligram (N=6) | BI 836826 25 Milligram (N=6) | BI 836826 50 Milligram (N=3) | BI 836826 100 Milligram (N=3) | BI 836826 200 Milligram (N=6) | BI 836826 400 Milligram (N=3) | BI 836826 800 Milligram (N=4)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cryptococcosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection fungal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 836826 1 Milligram (N=3) | BI 836826 3 Milligram (N=3) | BI 836826 9 Milligram (N=6) | BI 836826 25 Milligram (N=6) | BI 836826 50 Milligram (N=3) | BI 836826 100 Milligram (N=3) | BI 836826 200 Milligram (N=6) | BI 836826 400 Milligram (N=3) | BI 836826 800 Milligram (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 4 | 3 | 1 | 3 | 2 | 1 | 2
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 3 | 1 | 2 | 3 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 1 | 1 | 1 | 2 | 2 | 3
Aortic valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mitral valve calcification (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 3 | 2 | 2 | 0 | 2 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 3 | 3 | 0 | 1 | 2 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Submaxillary gland enlargement (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3 | 2 | 0 | 1 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 2 | 3 | 0 | 0 | 3 | 0 | 1
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 2 | 2 | 3 | 3 | 2 | 2 | 4 | 2 | 3
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Extravasation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Feeling of body temperature change (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 2 | 0 | 0 | 1 | 3 | 0 | 0
Puncture site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 4 | 3 | 2 | 2 | 3 | 1 | 2
Temperature regulation disorder (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug administration error (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 4 | 2 | 2 | 5 | 3 | 4
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure systolic increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Immunoglobulins decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
T-lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitamin B12 increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
pH urine decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 3 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Thrombosis in device (Product Issues) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 3 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 1
Pallor (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The trial was discontinued due to lack of recruitment before a formal maximum tolerated dose (MTD) was established based on the number of patients with Dose Limiting Toxicities (DLTs) in the first treatment cycle.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-10-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT01296932/SAP_000.pdf
  • Study Protocol (2015-03-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT01296932/Prot_001.pdf